CLINICAL TRIAL: NCT05859997
Title: A Clinical Study on the Safety and Efficacy of Universal CAR-T Cells (BRL-301) in the Treatment of Relapse or Refractory Autoimmune Diseases
Brief Title: Universal CAR-T Cells (BRL-301) in Relapse or Refractory Autoimmune Diseases
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Bioray Laboratories (Industry)
Collaborators: Shanghai Changzheng Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2022-BRL-301A-ADS-IIT
Record Dates: First submitted 2023-04-19; First posted 2023-05-16 (Actual); Last update posted 2024-11-20 (Actual); Status verified 2024-11

CONDITIONS: Systemic Lupus Erythematosus (SLE); Sjogren's Syndrome; Systemic Sclerosis; Inflammatory Myopathy; ANCA Associated Systemic Vasculitis; Antiphospholipid Syndrome
MeSH Terms: conditions — Lupus Erythematosus, Systemic; Sjogren's Syndrome; Scleroderma, Systemic; Myositis; Antiphospholipid Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- BRL-301 (Experimental): Allogeneic CD19-targeted Chimeric Antigen Receptor (CAR) T Cells
  Interventions: Biological: BRL-301

INTERVENTIONS:
Biological: BRL-301 — Single dose of Allogeneic Anti-CD19 CAR T cells will be infused
  Other Names: Allogeneic Anti-CD19 CAR T cells

SUMMARY:
This is an investigator initiated trial to assess the efficacy and safety of BRL-301 in the relapse or refractory autoimmune diseases of China.

DETAILED DESCRIPTION:
This is an investigator initiated trial to assess the efficacy and safety of BRL-301 in the relapse or refractory autoimmune diseases of China.

The study had the following sequential phases: Screening, Pre-Treatment (Cell Product Preparation & Lymphodepleting Chemotherapy), Treatment and Follow-up.

ELIGIBILITY:
Common Inclusion Criteria:

* Age ranges from 18 to 65 years old (including threshold), regardless of gender.
* Positive expression of CD19 on peripheral blood B cells determined by flow cytometry.
* The functions of important organs meet the following requirements:

  1. Bone marrow hematopoietic function needs to meet: a. White blood cell count ≥ 3 x 10^9/L b. Neutrophil count ≥ 1 x 10^9/L (no colony-stimulating factor treatment within 2 weeks before examination); c. Hemoglobin ≥60g/L.
  2. Liver function:ALT ≤ 3 x ULN,AST≤3 x ULN, TBIL≤1.5 x ULN(excluding Gilbert syndrome, total bilirubin ≤ 3.0 x ULN) (No requirements for conditions caused by the disease itself).
  3. Renal function: creatinine clearance rate (CrCl) ≥ 60 ml/minute(Cockcroft/Fault formula).
  4. Coagulation function: International standardized ratio (INR) < 1.5 x ULN,prothrombin time(PT) < 1.5 x ULN.
  5. Cardiac function: Good hemodynamic stability.
* Female subjects with fertility and male subjects whose partners are women of childbearing age are required to use medically approved contraception or abstinence during the study treatment period and at least 6 months after the end ofthe study treatment period; Female subjects of childbearing age tested negative for serum HCG within 7 days before enrollment in the study and were not in lactation.
* Voluntarily participate in this clinical study, sign an informed consent form, have good compliance, and cooperate with follow-up.

Criteria for SLE:

* Complies with the classification standards of the 2019 European Union Against Rheumatology/American Society of Rheumatology (EULAR/ACR) SLE.
* In the moderate to severe active phase of the disease, with SLEDAI-2000 score>6.
* And at least one British Isle Lupus Rating Group Index (BILAG-2004) Class A (severe manifestation) or two Class B (moderate manifestation) organ scores, or both.
* Ineffective conventional treatment or relapse of disease activity after remission. Definition of routine treatment: Use of glucocorticoids (above 1mg/Kg/d) and cyclophosphamide, as well as any of the following immunomodulatory drugs for more than 6 months: antimalarial drugs, azathioprine, mycophenolate mofetil, methotrexate, leflunomide, tacrolimus, cyclosporine, as well as biological agents such as rituximab, belimumab and telitacicept.

Criteria for Sjogren's syndrome with thrombocytopenia:

* Meets the 2002 AECG criteria for primary Sjogren's syndrome or the 2016 ACR/EULAR classification criteria.
* Diagnosed pSS-TP, platelet count < 30 × 10^9/L.
* Ineffective conventional treatment or relapse of disease activity after remission. Definition of routine treatment: Use of glucocorticoids (above 1mg/Kg/d) and cyclophosphamide, as well as any of the following immunomodulatory drugs for more than 6 months: antimalarial drugs, azathioprine, mycophenolate mofetil, methotrexate, leflunomide, tacrolimus, cyclosporine, as well as biological agents such as rituximab and belimumab.

Criteria for Systemic Sclerosis:

* Meets the classification criteria for Systemic Sclerosis according to the 2013 ACR, and conforms to diffuse manifestations.
* Concomitant interstitial pneumonia: interstitial changes with ground glass like exudate detected by chest HRCT.
* Needs to be met 1. or 2.:

  1. Ineffective conventional treatment or relapse of disease activity after remission. Definition of routine treatment: Use of glucocorticoids (above 0.5mg/Kg/d) and cyclophosphamide, as well as any of the following immunomodulatory drugs for more than 6 months: antimalarial drugs, azathioprine, mycophenolate mofetil, methotrexate, leflunomide, tacrolimus, cyclosporine, as well as biological agents such as rituximab and belimumab.
  2. Definition of progressiveness: a) Definition of skin progression: mRSS increases by>25%; b) The definition of lung disease progression: a 10% decrease in FVC, or a 5% decrease in FVC accompanied by a 15% decrease in DLCO.

Criteria for Inflammatory Myopathy:

* Classification criteria for inflammatory myopathy in accordance with 2017 EULAR/ACR (including DM, PM, ASS, and NM).
* For those with muscle involvement, the MMT-8 score is lower than 142 and at least two abnormalities are found in the following five core measurements (PhGA, PtGA, or extramuscular disease activity score ≥ 2 points; total HAQ score ≥ 0.25; muscle enzyme levels are 1.5 times the upper limit of the normal range).
* Myositis antibody positive.
* Needs to be met 1.or 2.:

  1. Ineffective conventional treatment or relapse of disease activity after remission. Definition of routine treatment: Use of glucocorticoids (above 1mg/Kg/d) and cyclophosphamide, as well as any of the following immunomodulatory drugs for more than 6 months: antimalarial drugs, azathioprine, mycophenolate mofetil, methotrexate, leflunomide, tacrolimus, cyclosporine, as well as biological agents such as rituximab and belimumab.
  2. Progressive definition: rapid progression of interstitial pneumonia in a short period of time.

Criteria for ANCA Associated Vasculitis:

* Meets the diagnostic criteria for ANCA vasculitis in 2022 ACR/EULAR, including microscopic polyangitis, granulomatous polyangitis, and eosinophilic granulomatous polyangitis.
* Positive ANCA related antibodies (MPO-ANCA or PR3-ANCA positive).
* The Birmingham Vasculitis Activity Scale (BVAS) is ≥ 15 points (a total score of 63 points), indicating the activity of the vasculitis condition.
* There must be at least one main item, at least three secondary items, or at least two renal items, hematuria and proteinuria, in the BVAS evaluation.
* Ineffective conventional treatment or relapse of disease activity after remission. Definition of routine treatment: Use of glucocorticoids (above 1mg/Kg/d) and cyclophosphamide, as well as any of the following immunomodulatory drugs for more than 6 months: antimalarial drugs, azathioprine, mycophenolate mofetil, methotrexate, leflunomide, tacrolimus, cyclosporine, as well as biological agents such as rituximab and belimumab.

Criteria for Antiphospholipid syndrome:

* Meets the diagnostic criteria for primary antiphospholipid syndrome revised in Sydney in 2006.
* Positive phospholipid antibodies with medium to high titers (IgG/IgM for LA, B2GP1, or acL, tested more than twice within 12 weeks).
* Needs to be met 1. or 2.:

  1. Use warfarin anticoagulation or replace the standard treatment of vitamin K antagonist (i.e. maintain the INR required for treatment) or use the standard treatment dose of low molecular weight heparin (LMWH), as well as use of hormones and cyclophosphamide to treat relapse thrombosis.
  2. Catastrophic antiphospholipid syndrome requires the following four criteria: (1) involving three or more organs, systems, and/or tissues; (2) Symptoms appear within 1 week; (3) Histologically confirmed obstruction of small blood vessels in at least one organ or tissue; (4) APL positive.

Exclusion Criteria:

* Individuals with a history of severe drug allergies or allergic constitution.
* Existence or suspicion of uncontrollable or treatable fungal, bacterial, viral or other infections.
* Individuals with relatively serious heart diseases, such as angina pectoris, myocardial infarction, heart failure, and arrhythmia.
* Subjects with congenital immunoglobulin deficiency.
* Other malignant tumors (excluding non-melanoma skin cancer, cervical cancer in situ, bladder cancer and breast cancer that have survived for more than 5 years without disease).
* Subjects with end-stage renal failure.
* Subjects with positive hepatitis B surface antigen (HBsAg) or hepatitis B core antibody (HBcAb) and HBV DNA titer in peripheral blood higher than the upper limit of detection; Patients with positive hepatitis C virus (HCV) antibodies and positive peripheral blood HCV RNA; People who are positive for human immunodeficiency virus (HIV) antibodies; Those who have tested positive for syphilis.
* Having mental illness and severe cognitive impairment.
* Those who have participated in other clinical trials within the first 3 months of enrollment.
* Pregnant or intending to conceive women.
* The researchers believe that there are other reasons why subjects cannot be included in this study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2023-05-17 (Actual); Primary Completion 2024-05-27 (Actual); Study Completion 2025-05-27 (Estimated)

PRIMARY OUTCOMES:
Safety and efficacy outcomes | First 30 days for DLT, 3 months for safety and efficacy measurements during the treatment assessment period, and then follow-up every 3 months for up to a year after the treatment.
  Safety assessments are conducted using the NCI-CTCAE version 5.0 standards；Efficacy assessments: Relapsed refractory systemic lupus erythematosus-SLE Response Index 4 (SRI-4) response;Sjögren's Syndrome with relapsed refractory thrombocytopenia-assessment of treatment response for thrombocytopenia(CR, PR, NR);Relapsed refractory/progressive systemic sclerosis-Composite Response Index in Systemic Sclerosis(CRISS);Relapsed refractory/progressive inflammatory myopathy-Total Improvement Score (TIS);Relapsed refractory ANCA-associated vasculitis-BVAS score;Recurrent Refractory/Catastrophic Antiphospholipid Syndrome-new thrombosis

SECONDARY OUTCOMES:
PK parameters | 3 months
  Changes in the CAR gene copy number and CAR-T cell count in peripheral blood and duration after infusion of BRL-301; time to peak (Tmax), peak concentration (Cmax), area under the concentration-time curve from 0 to 1 month (AUC0-M1), and from 0 to 3 months (AUC0-M3)
PD parameters | 3 months
  Changes in cytokines in peripheral blood after infusion of BRL-301

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai ChangZheng hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Wang D, Wang X, Tan B, Wen X, Ye S, Wu Y, Cao X, Zhang X, Wang C, Geng L, Zhang H, Feng X, Zheng B, He Y, Liu M, Wu X, Du B, Sun L, Xu H. Allogeneic CD19-targeted CAR-T therapy in refractory systemic lupus erythematosus achieved durable remission. Med. 2025 Oct 10;6(10):100749. doi: 10.1016/j.medj.2025.100749. Epub 2025 May 29. PMID 40446794
- [Derived] Wang X, Wu X, Tan B, Zhu L, Zhang Y, Lin L, Xiao Y, Sun A, Wan X, Liu S, Liu Y, Ta N, Zhang H, Song J, Li T, Zhou L, Yin J, Ye L, Lu H, Hong J, Cheng H, Wang P, Li W, Chen J, Zhang J, Luo J, Huang M, Guo L, Pan X, Jin Y, Ye W, Dai L, Zhu J, Sun L, Zheng B, Li D, He Y, Liu M, Wu H, Du B, Xu H. Allogeneic CD19-targeted CAR-T therapy in patients with severe myositis and systemic sclerosis. Cell. 2024 Sep 5;187(18):4890-4904.e9. doi: 10.1016/j.cell.2024.06.027. Epub 2024 Jul 15. PMID 39013470